CLINICAL TRIAL: NCT06825039
Title: The Effects of Extracorporeal Shock Wave Therapy in Different Stages of Scar Formation in Postsurgical Scars Especially After Abdominplasty and Breast Reduction.
Brief Title: The Effects of Extracorporeal Shock Wave Therapy in Postsurgical Scars Especially After Abdominplasty and Breast Reduction.
Acronym: Effect of SWT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Heilig Hart Ziekenhuis Lier (Unknown); University Hospital, Antwerp (Other); Ziekenhuis Rivierenland (Other); AZ Middelheim, Antwerpen (Unknown)
Responsible Party: Principal Investigator, Ulrike Van Daele, Principal Investigator, Universiteit Antwerpen
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11B8619N(BELGIUM); 2613 (Other: University of Antwerp)
Record Dates: First submitted 2024-12-16; First posted 2025-02-13 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Scar; Shockwave Therapy
Keywords: Skin scars, Post surgical, Underlying mechanisms, Shock wave
MeSH Terms: conditions — Cicatrix | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Focused ESWT will be applied to the scarred area in the 3 intervention groups. Each group will receive 10 ESWT treatments with a frequency of 1x/week. Energy levels (EFD mJ/mm2) or bar in radial can range between 0.01-0.33 mJ/mm2. Based upon experimental papers, the described energy flux density, frequency and number of shots should activate or modulate the signaling pathways of interest and are used in the treatment of scars.
  Concept of low-energy treatments for group 3 (ESWT 1) and 4 (ESWT 2):
  * Intensity: 0.07mJ/mm2
  * Number of shocks: 100 impulses/cm2
  * Frequency: 2 Hz
  * Treatment frequency: 1x/week
  * Total amount of treatments: 10 treatments
  Concept of high-energy treatments for group 5 (ESWT 3):
  * Intensity: 0.25mJ/mm2
  * Number of shocks: 100 impulses/cm2
  * Frequency: 8 Hz
  * Treatment frequency: 1x/week
  * Total amount of treatments: 10 treatments The scarred area is prepared with contact-gel to conduct the shock waves. The investigators treat scars after full wound closure.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 3 (Experimental): * Intensity: 0.07mJ/mm2
  * Number of shocks: 100 impulses/cm2
  * Frequency: 2 Hz
  * Treatment frequency: 1x/week
  * Total amount of treatments: 10 treatments
  Interventions: Device: Shockwave therapy
- Group 5 (Experimental): * Intensity: 0.25mJ/mm2
  * Number of shocks: 100 impulses/cm2
  * Frequency: 8 Hz
  * Treatment frequency: 1x/week
  * Total amount of treatments: 10 treatments
  Interventions: Device: Shockwave therapy
- Group 1 (No Intervention): Control group
- Group 2 (No Intervention): Control group
- Group 4 (Experimental): * Intensity: 0.07mJ/mm2
  * Number of shocks: 100 impulses/cm2
  * Frequency: 2 Hz
  * Treatment frequency: 1x/week
  * Total amount of treatments: 10 treatments
  Interventions: Device: Shockwave therapy

INTERVENTIONS:
Device: Shockwave therapy — Focused ESWT will be applied to the scarred area in the 3 intervention groups. Each group will receive 10 ESWT treatments with a frequency of 1x/week. Energy levels (EFD mJ/mm2) or bar in radial can range between 0.01-0.33 mJ/mm2 (33). Based upon experimental papers, the described energy flux density, frequency and number of shots should activate or modulate the signaling pathways of interest and are used in the treatment of scars.
  Arms: Group 3; Group 4; Group 5

SUMMARY:
Scars can be caused by physical trauma, surgical incisions, burn injuries and even acne. Deep cutaneous injuries induce pathological scars. Other factors, such as mechanical loading, bacterial colonization are potential factors thought to underlie human hypertrophic and keloid scar formation or contractures. The effect may include functional impairment and aesthetic disadvantages.

Various non-invasive mechanical interventions of physical scar management (e.g. extracorporeal shock wave therapy or ESWT) could have a beneficial influence on wound healing and prevention of hypertrophic scars. ESWT considerably improves the appearance and symptoms of hypertrophic scars. However, the mechanism underlying the observed beneficial effects is not well understood. The objective of the first part of the study is to elucidate the mechanism underlying changes in cellular mechanosensitive pathways that are induced by ESWT. This review will introduce the histopathological effects on ESWT during wound healing and scar development.

The main objective of this study is to determine how much mechanical loading on dermal scars will lead to normal scar healing. The optimal duration, the frequency and the intensity of the applied forces in ESWT to generate a beneficiary effect during different phases of wound healing remains unclear.

In this study, biopsies from abdomionplasty postsurgical scars will be examined. Thereby it is possible to evaluate the outcomes on a cellular level through assessing the histology of human biopsies under controlled condition. In the second part, the underlying mechanism of ESWT on postsurgical scars will be explored, in different stages of wound healing. Furthermore, the investigators will investigate if changes in physical characteristics (redness, thickness and pliability) in postsurgical scars are associated with changes in reactivity of mechanosensitive pathways. This study will close the gap between the fundamental knowledge on cellular mechanotransduction and the clinical application of mechanotherapy during physical scar management (ESWT).

DETAILED DESCRIPTION:
1. State of the art Every year 80 million scars develop in the world and 40-70% of these will develop into hypertrophic or problematic scars. Moreover, fibrosis and scar formation of the skin pose a substantial physiological and psychological burden on patients. Scars can be caused by physical trauma, surgical incisions, burn injuries and even acne. Most superficial injuries, that do not reach the dermis, do not leave significant scars. However, deep cutaneous injuries can induce pathological scars. Such scars often result in pain, itching, functional impairment, aesthetic disadvantages, anxiety, depression and poor quality of life of the affected person. All these aspects may cause poor functioning during ADL (4). Other aspects, such as uncontrolled mechanical loading, prolonged inflammation, overactive proliferation, bacterial colonization, and foreign-body reaction are potential factors thought to underlie human hypertrophic and keloid scar formation or contractures.

   Recent studies have identified that under influence of mechanical load scar proliferation will be prolonged and will even prohibit full maturation of the scar within the foreseen timeframe of two years of wound healing. Mechanical loading can be regarded as any mechanical stress applied to a healing wound, for example imposed forces during physical therapy or tensile forces during activities of daily living. It has been proven that specific sites that are frequently subjected to mechanical load during daily activities have more risk to develop into hypertrophic scars.

   Interestingly, mechanical loading cannot only be regarded as a negative predictive factor in scar formation. Under controlled conditions, mechanical load can activate a process called 'mechanotransduction'. Once activated inflammation, proliferation and thereby fibrosis and hypertrophic scarring can be regulated/controlled. Thus, mechanotransduction can be defined as the intracellular conversion of mechanical stimuli into internal chemical signals resulting in gene transcription. This has an effect on the cytoskeleton and the ECM. Signaling pathways are activated or modulated resulting in modification of the affected (scar) tissue.

   Various non-invasive mechanical interventions of physical scar management (e.g. extracorporeal shock wave therapy or ESWT, pressure therapy, vacuum massage,..) apply mechanical load and thereby initiate mechanotransduction. Controlled physical scar management can have a beneficial influence on wound healing and prevention of pathological scars. Therefore, this study will focus on the application of mechanical forces in the form of ESWT application. ESWT considerably improves the appearance and symptoms of hypertrophic scars. However, the mechanisms underlying the observed beneficial effects in scar management is not well understood.

   To date, there is no consensus concerning the optimal standard of care in scar treatment. Therefore, there is a need to study the underlying mechanism of scarring and the related influence of controlled mechanical forces.
2. Rationale of the study The heterogeneity in causes of scars, the complicated histology of scarring and the numerous intervention possibilities make late-stage clinical research in this field a search for a needle in a haystack. Moreover, it is always difficult to control variables such as location, demographics and genetics in studies.

First, proper identification of the cause and scar type is necessary to understand the complicated pathophysiology of excessive scarring. In this study, human dermal scar biopsies from patients who had undergone an abdominoplasty will be examined. By focusing on one specific region and one type of surgery, the influence of localization in wound healing will be controlled and a more homogenous scar formation process can be expected.

Abdominoplasty is one of the most frequently performed procedures in aesthetic surgery making that subjects can be more readily recruited and tested. An abdominoplasty is performed for various reasons: bariatric patients after weight loss with residual excess skin, post pregnancy patients to restore their previous appearance and the aging population who wants to maintain their youth belly. It's general aim is to remove the excess skin and fat, as well as to tighten the abdominal muscle. A surgeon will try to perform this procedure with the smallest possible incision. To ensure the best possible postsurgical scar outcome, preoperative incision planning, wound tension during closure, and postsurgical management (e.g. postsurgical dressing) are all critical. After an abdominoplasty, patients get the advice to use a scar cream, silicone tape and scar massage. However, as mentioned earlier surgical scars could result in contracting scars from a hypertrophic scar.

Currently, animal models (mice, pig and rabbit ear) are mostly used to unravel the pathophysiology of scarring and to develop new therapies. Underlying mechanisms in fibrosis research is heavily reliant on in vivo animal models, due to ethical and logistical limitations. Because of ethical concerns most human studies on the underlying mechanism of scars, have been limited to observational studies.

Unfortunately, animal models aren't able to reproduce the normal process of hypertrophic scar development as occurs in humans. For example, in murine models, the resting tension of the skin is lower in human skin. In addition, laboratory animals have a fibromuscular layer under the dermis, which is considered to be the main pathological difference to humans.

Skin biopsies provide valuable information on cellular and molecular level of a human dermal scar. Because of the accessibility of the skin and application of local anaesthesia, skin biopsies can be performed quite easy. By assessing the histopathology of human dermal skin biopsies the investigators will be able to study the mechanism under controlled conditions and evaluate the outcome on a cellular and molecular level. In addition, the overall cosmetic result of a punch biopsy is well-accepted and has a low complication and infection risk. Furthermore, patients after an abdominoplasty have an incision that is approximately 75 cm long making it possible to obtain a biopsy for our study.

There are some preliminary studies that took a biopsy in human dermal scars to examine the cellular and molecular changes. In vivo patient scarring research, by examining human dermal skin biopsies, enables us to study scar pathogenesis and thereby effect of therapeutic scar treatment. This kind of research is, to the best of our knowledge, the most representative model for the underlying mechanism of human wound healing and scarring.

In this study, the investigators will investigate one intervention, namely ESWT. ESWT meets all the requirements for the ideal scar treatment. ESWT is a non-invasive scar treatment, well tolerated by patients, easy to apply and it has a precise control of load intensity and frequency. In addition, it has low complication rates and is easy to use in outpatient settings. ESWT is also cost-effective and can already be applied during wound healing and early scar formation and thus can be used as a preventive therapy for pathological scars.

Only a few studies have examined the effects of ESWT in combination with surgical techniques. Preliminary results showed that ESWT diminishes the adverse effects of the surgical procedure and wound healing can be improved. An increased perfusion and angiogenesis in the wound due to increased systemic growth factor expression are thought to be responsible this effect. Finally, the application of ESWT, post-surgery, has also beneficial clinical results for the patients. Studies demonstrate that all relevant physical and physiological scar parameters such as height, pliability, vascularity and pigmentation, improve after ESWT. These changes will ameliorate function, which is, among others, demonstrated on retracting hand scars by an increase of passive ROM. From this previous research the investigators can conclude that it is safe to apply ESWT after surgery. Only one study was found on ESWT by abdominoplasty. This pilot study examined the effect of preoperative ESWT on the postoperative scar formation. Patients who had undergone and abdominoplasty were conducted and were preoperatively allocated to low energy ESWT or placebo. Scar formation was evaluated by 19 different scar parameters. This study showed that ESWT reduces scar formation and postoperative symptoms after abdominoplasty surgery. The largest differences were observed in thickness and overall impression of the scar (Vancouver scar scale). Together with other ESWT research the investigators therefore hypothesize: that postoperative ESWT have beneficial effects after abdominoplasty surgery. As it is already proven preoperative, ESWT application after surgery presumably have advantages on quality of life and reduce pain.

This study will close the gap between the fundamental knowledge on mechanotransduction and the clinical application of mechanotherapy during physical scar management (especially ESWT) by:

1. examining the association of the cellular and molecular changes with the changes in physical characteristics of scars
2. using different treatment modalities in ESWT
3. during different wound healing phases

Although some studies have been performed on ESWT for prevention of hypertrophic and keloid scars, the exact mechanism remains largely unclear. Based upon current clinical research the optimal duration, the frequency and the energy levels of the applied forces in ESWT to generate a beneficiary effect on scar formation remain unclear. Furthermore, it has not yet been proven that there is an association between these mechanosignaling pathways and physical and physiological changes during different phases in scar formation. This study will be the stepping stone towards future late stage clinical research in non-invasive scar management.

Novelty in this study:

* standardizable: 1 type and location of surgery scar: scar after abdominoplasty
* controllable load application: extracorporeal shock wave therapy or ESWT
* evaluation of the outcome on different levels:

  1. cellular and molecular through assessing the histopathology and molecular mechanosignaling pathways.
  2. scar level through physical non-invasive scar assessments (thickness, elasticity, and colour of the scar).

  3. Research objectives In this study the investigators will elucidate the mechanisms underlying changes in cellular and molecular mechanosensitive pathways that are induced by ESWT. More specifically, in this study, changes in amount of ∝-SMA, myofibroblast, macrophages, TGF-β, collagen, TLR3, collagen orientation and the angiogenetic process will be examined. Furthermore, the investigators want to determine how much mechanical loading on dermal scars will lead to normal scar healing. In addition, physical outcomes will be measured by subjective and objective assessments.

The underlying mechanism of the application of ESWT on postsurgical scars will be explored, in different stages of wound healing by taking a biopsy before and after treatment and at a fixed time during scar formation. A control group (without ESWT treatment) will be compared with an intervention group (with ESWT treatment). In the intervention group different ESWT modalities will be applied, during different stages scar formation (especially during the proliferation and maturation phase). Besides, the investigators will investigate if changes in physical characteristics (pain, colour, thickness, pliability and quality of life) in postsurgical scars are associated with changes in reactivity of mechanosensitive pathways in the different control or intervention group during different stages of scar formation.

ELIGIBILITY:
Inclusion criteria

* Eligible patients aged between 18 and 80 years
* Dutch or English speaking
* Patients who had undergone an abdominoplasty resulting in a dermal scar
* Informed consent (approved by the ethics committee) will be provided before the surgical intervention Exclusion criteria
* All type of skin diseases or dermatological problems
* Previous surgery or ESWT intervention at the current scar site
* Age under 18 years or above 80 years
* Inability to provide informed consent
* Expected problems in therapy compliance or follow up
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in α-SMA and myofibroblasts | baseline: 2weeks and 6 weeks OR 6 weeks and 3 weeks
  Scar tissue biopsy specimens will be collected by an experienced plastic surgeon from patients who had undergone an abdominoplasty that registered for the study. The biopsy will be embedded in paraffin for histological examination. After application of local anaesthesia, a 3-4mm diameter punch biopsy will be taken to ensure the presence of the subcutis in the biopsy and to ensure sufficient tissue. After the biopsy has been taken, the small lesion will be closed by a single suture.
  The investigators are interested in change in α-SMA and myofibroblasts by immunohistochemistry.
Change in Macrophages | baseline: 2weeks and 6 weeks OR 6 weeks and 3 weeks
  Scar tissue biopsy specimens will be collected by an experienced plastic surgeon from patients who had undergone an abdominoplasty that registered for the study. The biopsy will be embedded in paraffin for histological examination. After application of local anaesthesia, a 3-4mm diameter punch biopsy will be taken to ensure the presence of the subcutis in the biopsy and to ensure sufficient tissue. After the biopsy has been taken, the small lesion will be closed by a single suture. The investigators are interested in change in macrophages by immunohistochemistry.
Change in TGF-β | baseline: 2weeks and 6 weeks OR 6 weeks and 3 weeks
  Scar tissue biopsy specimens will be collected by an experienced plastic surgeon from patients who had undergone an abdominoplasty that registered for the study. The biopsy will be embedded in paraffin for histological examination. After application of local anaesthesia, a 3-4mm diameter punch biopsy will be taken to ensure the presence of the subcutis in the biopsy and to ensure sufficient tissue. After the biopsy has been taken, the small lesion will be closed by a single suture. The investigators are interested in change in TLR3 by immunohistochemistry.
Change in collagen type I en type III | baseline: 2weeks and 6 weeks OR 6 weeks and 3 weeks
  Scar tissue biopsy specimens will be collected by an experienced plastic surgeon from patients who had undergone an abdominoplasty that registered for the study. The biopsy will be embedded in paraffin for histological examination. After application of local anaesthesia, a 3-4mm diameter punch biopsy will be taken to ensure the presence of the subcutis in the biopsy and to ensure sufficient tissue. After the biopsy has been taken, the small lesion will be closed by a single suture. The investigators are interested in change in collagen type I en type III by immunohistochemistry.

SECONDARY OUTCOMES:
Measurement of color changes in scar tissue | baseline: 2 weeks - 6 weeks - 3 months - 6 months
  Colour will be measured using a Mexameter MX18 (from Courage and Khazaka) using the erythema/melanin indices. The Mexameter uses 16 light-emitting diodes that emit light at three wavelengths (green: 568 nm; red 660 nm; infrared 880 nm). Then, the reflected light is measured by a receiver unit. Erythema is measured by the green and red wavelengths, whereas melanin is determined by the red and infrared wavelengths.
Measurement of vertical elasticity changes in scar tissue | baseline: 2 weeks - 6 weeks - 3 months - 6 months
  Vertical elasticity will be measured using a Cutometer Dual MPA 580®(from Courage and Khazaka). The cutometer uses a negative pressure where after the skin is drawn into the aperture of the probe.
Patient-reported outcomes on scar characteristics | baseline: 2 weeks - 6 weeks - 3 months - 6 months - 1 year
  The patient observer scar assessment scale is a two numerical scar assessment scale whereby the patient and observer evaluate the scar.
  The observer scar assessment scale-observer scale (POSAS-O 3.0) is filled in by the investigator. POSAS-P 3.0 (patient) is filled in by the patient and is a reliable instrument. A total of 16 or 17 items in the generic and linear questionnaire, aimed at measuring visual (e.g., color), tactile (e.g., pliability), and sensory (e.g., itching) characteristics of the scar. Additionally, there is 1 item regarding overall satisfaction with the scar (this item is excluded from the scoring). Each item is rated on a scale from 0 to 10, where 0 represents the best possible outcome (no scar or no issues) and 10 represents the worst possible outcome (severe issues with the scar).
Quality of life assessment in scar-affected Individuals | baseline: 2 weeks - 6 weeks - 3 months - 6 months - 1 year
  The Dermatology Life Quality Index (DLQI) is a questionnaire to define patient satisfaction. It quantifies the health-related quality of life of the patient by measuring the disability caused by any skin disease.
  The DLQI consists of 10 questions, each addressing a different aspect of how the skin condition affects the patient's life. Each question is scored on a scale from 0 to 3, where: 0 = "Not at all" (no impact); 1 = "A little" (small impact); 2 = "A lot" (moderate to significant impact); 3 = "Very much" (severe impact). The maximum possible score is 30 (if all answers are "3"). The minimum possible score is 0 (if all answers are "0").
  Interpreting the DLQI Score:
  0-1: No effect on quality of life 2-5: Small effect on quality of life 6-10: Moderate effect on quality of life 11-20: Very large effect on quality of life 21-30: Extremely large effect on quality of life
Quality of life assessment in scar-affected Individuals | baseline: 2 weeks - 6 weeks - 3 months - 6 months - 1 year
  EQ-5D-5L includes items on five domains. Mobility/ Self-care/ Usual activities/pain, discomfort/ Anxiety / Depression/EQ overall haelth assessed on a Visual Analogue Scale.
  Scoring System of the EQ-5D-5L:
  Each of the 5 dimensions is scored on a 5-level scale (from 1 to 5), where:
  1. = No problems
  2. = Slight problems
  3. = Moderate problems
  4. = Severe problems
  5. = Extreme problems ) These responses are used to calculate a health state that is mapped to an index score ranging from 0 (worst health) to 1 (best health), reflecting overall health status. Additionally, a Visual Analog Scale (VAS) allows individuals to rate their perceived health on a scale from 0 (worst health) to 100 (best health).

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - Ziekenhuis aan de Stroom, Antwerp, Antwerp
  - Heilig Hart Ziekenhuis Lier, Lier, Antwerp
  - AZ Rivierenland Rumst, Rumst, Antwerp
  - Universitair Ziekenhuis, Wilrijk, Antwerp

IPD SHARING:
Plan to Share IPD: No
Datasets will be made available upon request.